CLINICAL TRIAL: NCT06456515
Title: A Single-Arm, Multicenter Phase II Clinical Study of Regorafenib and Sintilimab in Combination with Electroacupuncture in Patients with MSS Advanced Colorectal Cancer Who Have Failed More Than Second-Line Standard Chemotherapy
Brief Title: Regorafenib and Sintilimab in Combination with Electroacupuncture in MSS CRC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Principal Investigator, Wenwei Hu, Vice Director of Oncology Department, The First People's Hospital of Changzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-IRB-SOP-00710
Record Dates: First submitted 2024-05-21; First posted 2024-06-13 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Regorafenib; Sintilimab; electroacupuncture; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; sintilimab; Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Regorafenib and Sintilimab in combination with electroacupuncture (Experimental)
  Interventions: Drug: Regorafenib and Sintilimab in combination with electroacupuncture

INTERVENTIONS:
Drug: Regorafenib and Sintilimab in combination with electroacupuncture — Regorafenib, take for 2 weeks and stop for 1 week; Sintilimab, intravenous, every 3 weeks; Electroacupuncture was performed 1 day before, on the day of, and on the 2nd day after each cycle of Sintilimab administration, and patients completed 3 treatments in week 1, followed by 1 treatment per week for 2 weeks, with 5 treatments per dosing cycle.

SUMMARY:
The aim of this clinical trial is to find out whether Regorafenib and Sintilimab in combination with electroacupuncture works in treating participants with microsatellite stable (MSS) advanced colorectal cancer who have failed one or more second-line standard chemotherapy regimens. It will also learn about the efficacy and safety of the combination therapy. The main questions the trial aims to answer are:

Does combination therapy reduce the overall survival time ? What medical problems do people have when they take combination therapy?

Participants will

Regorafenib, take for 2 weeks and stop for 1 week; Sintilimab, intravenous, every 3 weeks; Electroacupuncture was performed 1 day before, on the day of, and on the 2nd day after each cycle of Sintilimab administration, and patients completed 3 treatments in week 1, followed by 1 treatment per week for 2 weeks, with 5 treatments per dosing

ELIGIBILITY:
Inclusion Criteria:

1. Fullly knowledge of the study and voluntarily sign the informed consent;
2. Histologically and/or cytologically confirmed metastatic colorectal adenocarcinoma (Stage IV) with microsatellite stable (MSS)* confirmed by PCR or NGS;
3. Receive at least two lines of standard chemotherapy in the past and have failed.
4. No systemic chemotherapy or antitumor therapy such as radiotherapy, immunotherapy, biological or hormonal therapy in the past 4 weeks; and have never received VEGFR inhibitors
5. Willing to receive electroacupuncture;
6. Aged 18-75 years old (including 18 years old and 75 years old);
7. Weighing more than 40 kg (including 40 kg);
8. Able to take oral medication.
9. Patients with adequate organ function at the time of enrollment are defined as follows: Neutrophil count ≥1500mm3 Platelet count ≥10.0 × 104/mm3 Hemoglobin (Hb) ≥ 9 g/dL Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤100 U/L (≤100 U/L in patients with hepatocellular carcinoma, ≤250 U/L in patients with liver metastasis) Total bilirubin ≤1.5 mg /dL Creatinine ≤1.5 mg /dL Lipase ≤ 80 IU/L Urine Protein: one of the following (if any of the criteria are met, no other test may be performed) (i) Urine Protein (paper test) of 2+ or less (ii) UPC < 3.5 (iii) Urine Protein ≦ 3500 mg for 24 hour urine protein measurements. mg Prothrombin time (PT)-International Normalized Ratio (INR): ≤ 1.5 (≤ 3.0 for anticoagulant administration)
10. Eastern Cooperative Oncology Group Physical Performance Score (ECOG PS) ≤ 1 (0-1);
11. Cardiac function evaluation: left ventricular ejection fraction ≥ 50% (echocardiography);
12. Clearly meet the criteria for evaluating the efficacy of solid tumors (e.g., echocardiograms) Measurable lesions that meet the requirements of RECIST 1.1;
13. Expected survival of more than 12 weeks.

Exclusion Criteria:

Patients will be excluded from the study if any of the following criteria are met.

1. Patients who have received systemic chemotherapy, radiotherapy, surgery, hormonal therapy or immunotherapy <2 weeks prior to enrolment. Immune checkpoint blockade pretreatment is permitted.
2. Patients with a history of regorafenib administration.
3. Patients with uncontrolled hypertension (systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥90 mmHg) despite multiple antihypertensive medications; and
4. Patients with acute coronary syndromes (including myocardial infarction and unstable angina) and a history of coronary angioplasty or stenting within 6 months prior to enrolment;
5. Patients with a large pleural effusion or ascites requiring drainage; and
6. Patients with grade ≥ 3 active infection according to NCI CTC AE version 4.03; patients with symptomatic brain metastases; and patients with a history of coronary artery angioplasty or stenting within the previous 6 months.
7. Patients with symptomatic brain metastases;
8. Patients with partial or complete gastrointestinal obstruction;
9. Patients with interstitial lung disease with active signs or symptoms;
10. Patients who test positive for anti-HIV-1 antibody, anti-HIV-2 antibody, hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (HCV)* *Patients who test positive for anti-hepatitis B surface (HBs) or anti-hepatitis B core (HBc) antibodies and patients with hepatitis B virus (HBV)-DNA measurements that are greater than the sensitivity of the test will also be excluded. Patients with concurrent autoimmune disease
11. Patients with concurrent autoimmune disease or a history of chronic or recurrent autoimmune disease.
12. Patients requiring systemic corticosteroids (excluding those given temporarily for testing, prophylactic administration for allergic reactions, or for the relief of swelling associated with radiotherapy) or immunosuppressive agents, or who have received such therapy <14 days prior to study participation;
13. Patients with a history or finding of class ≥III congestive heart failure according to the New York Heart Association functional class;
14. Patients with epilepsy requiring pharmacological treatment;
15. Patients with grade 3 or greater bleeding within 4 weeks prior to enrolment.
16. Patients who have undergone major surgery (open heart or caesarean section, etc.), caesarean biopsy, or trauma within 28 days prior to enrolment. the same day of the week prior to the 4-week period may be enrolled (however, in the case of manual anastomosis without bowel resection, this should be within 14 days prior to enrolment);
17. Patients with non-healing wounds, non-healing ulcers or non-healing fractures.
18. Patients with a history of hypersensitivity reaction to any investigational drug, analogue or excipient.
19. Women who are pregnant or breastfeeding or have the potential to become pregnant.
20. Patients with contraindications to electroacupuncture therapy or patients for whom electroacupuncture is contraindicated in accordance with TCM syndromes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 2 years
  The time from randomization to death

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  The proportion of patients that respond either partially or fully to therapy
Progression-free survival (PFS) | Up to 2 years
  The time from randomization until first evidence of disease progression or death
Disease control rate (DCR) | Up to 2 years
  Percentage of patients with advanced cancer whose therapeutic intervention has led to a complete response, partial response, or stable disease
Time to progression (TTP) | Up to 2 years
  The time from randomization until first evidence of disease progression
Health-related quality of life (HRQoL) | Up to 2 years
  Assessment of patient quality of life with respect to health status
Adverse events (AE) | Up to 2 years
  Use the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
  Overall incidence of TEAE;
  * Incidence of grade 3 or higher AE;
  * Incidence of SAEs;
  * Incidence of AEs leading to permanent discontinuation;
  * Incidence of AEs leading to medication suspension or dose adjustment.
Cancer-related fatigue(CRF) | Up to 2 years
  A distressing, persistent, subjective sense of physical, emotional, and/or cognitive tiredness or exhaustion related to cancer and/or cancer treatment that is not proportional to recent activity and interferes with usual functioning, use the Revised Piper Fatigue Scale (RPFS)
Biomarker | Up to 2 years
  Biomarker analysis can be categorized as "non-genetic" (e.g., associated proteins) or "genetically relevant" (e.g., associated RNA or DNA).
Cmax | Up to 2 years
  Based on non-compartmental PK evaluation.Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
  Blood samples should be collected within 2 hours before electroacupuncture administration and 1 to 4 hours after electroacupuncture by weeks 2 and 3, and 2 hours before electroacupuncture in cycles 4-6
Immune-related adverse event (irAE) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Changzhou, Changzhou, China